CLINICAL TRIAL: NCT06406699
Title: Feasibility and Acceptability of Group Pain Reprocessing Therapy for Veterans With Chronic Neck/Back Pain
Acronym: ESPRIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-1387
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Chronic Back Pain; Chronic Pain; Neck Pain; Back Pain
MeSH Terms: conditions — Chronic Pain; Neck Pain; Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pain Reprocessing Therapy (Experimental): Participants will participate in once weekly telehealth group pain reprocessing therapy. Sessions will last approximately 1 hour in length. Group size will be approximately 10 individuals.
  Interventions: Behavioral: Pain Reprocessing Therapy (PRT)

INTERVENTIONS:
Behavioral: Pain Reprocessing Therapy (PRT) — PRT is a psychological intervention for chronic pain patients with a primary nociplastic component. PRT aims to help patients reconceptualize their pain as a non-dangerous signal that is not indicative of tissue pathology or structural abnormality. Through decreasing the threat level of their chronic pain, the pain itself can also resolve.

SUMMARY:
The investigators are conducting a trial that evaluates the feasibility of telehealth group pain reprocessing therapy (PRT), with no comparison group, for the treatment of chronic back pain in a population of veterans. PRT is a psychotherapy for chronic pain that aims to help patients reconceptualize their pain as a non-dangerous signal. It has been shown to be effective in a previous RCT (n=151).

ELIGIBILITY:
Inclusion Criteria:

* At least 6 months of back pain with last week average back pain at least 4/10
* Able to attend at least 7/8 telehealth group sessions
* Access to safe living space, quite room, reliable internet, and electronic device that can be used to attend telehealth therapy sessions.

Exclusion Criteria:

* Leg pain that is worse than back pain
* Suicide attempt, SI, HI, or inpatient psychiatric hospitalization in the past 5 years
* Not receiving/has not received disability or workers compensation related to back pain in the past 2 years.
* Is not currently involved in litigation regarding chronic back pain.
* Current misuse or overuse of alcohol or drugs
* Major surgery or other major medical events in the next 6 months
* Known vertebral/spinal fracture or tumor.
* Back surgery within last 2 years
* Difficulty controlling bowel movements
* Current or recent diagnosis of cancer
* Current or recent diagnosis of severe cardiovascular disease
* Unexplained or unintended greater than 20 pound weight loss in the past year
* Diagnosis of rheumatoid arthritis, polymyalgia rheumatica, scleroderma, Lupus, polymyositis, or other specific inflammatory disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2024-04-17 (Actual); Primary Completion 2025-01-25 (Actual); Study Completion 2025-02-08 (Actual)

PRIMARY OUTCOMES:
PEG-3 Average Pain in last week | Baseline, Post-treatment, and 2-months post-treatment
  0-10 scale that asks participant to rate their average pain (0=No pain, 10=Pain as bad as possible) in the last week

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado - Anschutz Medical Campus VA, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No